CLINICAL TRIAL: NCT05898620
Title: A Baseline-Controlled, Open-Label, Multicenter, Single-Arm, Pivotal Study to Evaluate the Efficacy, Safety, and Tolerability of NGN-401 in Subjects With Rett Syndrome (Embolden)
Brief Title: A Novel, Regulated Gene Therapy (NGN-401) Study for Females With Rett Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurogene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RTT-200
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rett Syndrome
Keywords: Typical Rett Syndrome; MECP2; Rett Disorder; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Neurodevelopmental Disorders; Neurobehavioral Manifestations; Neurologic Manifestations; Intellectual Disability; Nervous System Diseases; Pathologic Processes; RTT
MeSH Terms: conditions — Rett Syndrome; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Neurodevelopmental Disorders; Neurobehavioral Manifestations; Neurologic Manifestations; Intellectual Disability; Nervous System Diseases; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: The study treatment will be delivered via intracerebroventricular (ICV) injection. All study participants will receive the same intervention.
Who Masked: Outcomes Assessor
Masking Description: Central raters for the acquisition of a developmental milestone/skill from videos are blinded to the intervention and to the timing of the video.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pediatric 1e15 vg dose (fully enrolled) (Experimental): Dose Level 1 for ages 4-10 years
  Interventions: Genetic: NGN-401
- Adolescent/Adult 1e15 vg Dose (fully enrolled) (Experimental): Dose Level 1 for ages 11 years & above
  Interventions: Genetic: NGN-401
- Pediatric 3e15 vg dose (discontinued) (Experimental): Dose Level 2 for ages 4-10 years (discontinued)
  Interventions: Genetic: NGN-401
- Pivotal Cohort (Experimental): Dose Level 1 for ages 3 and above
  Interventions: Genetic: NGN-401

INTERVENTIONS:
Genetic: NGN-401 — NGN-401 is a non-replicating, recombinant AAV9 carrying a full length human MECP2 transgene.

SUMMARY:
This study will evaluate the efficacy and safety profiles of the investigational gene therapy, NGN-401, in females with typical Rett syndrome.

DETAILED DESCRIPTION:
The pivotal study, Embolden (TM), is a conversion of the phase 1/2 study and is an open-label, baseline-controlled, multicenter, single-arm study designed to assess the efficacy, safety, and tolerability of administration of NGN401, an adeno-associated viral vector serotype 9 (AAV9) using Neurogene's proprietary transgene regulation technology. NGN-401 contains a full-length human MECP2 gene and is designed to express therapeutic levels of the MeCP2 protein while avoiding overexpression.

The study treatment will be given as a single administration under general anesthesia via intracerebroventricular (ICV) delivery. Each participant will be followed for efficacy and safety for 3 years after treatment, and is expected to enroll in a long-term follow-up study for 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Females who are between the ages of ≥4 and ≤10 years for Arms 1 and 2 (Arms closed). Females who are ≥11 years of age or older for Arm 3 (Arm closed). Females who are ≥3 for Arm 4, the pivotal cohort.
* Diagnosis of typical Rett syndrome with a documented disease-causing mutation in the methyl-CpG-binding protein 2 (MECP2) gene
* Current anti-epileptic drug regimen has been stable for at least 12 weeks
* Participant must be in the post-regression stage
* Participant and caregiver should reside within a 2-hour drive of the study center for at least 3 months following treatment
* Participant must have never taken trofinetide or have taken trofinetide and discontinued due to tolerability, lack of efficacy, or other reasons. Following NGN-401 dosing, trofinetide may be initiated after a specified time period and with the support of the treating clinician.

Exclusion Criteria:

* Normal or near normal hand function
* Has a current clinically significant condition other than Rett syndrome
* Presence of a concomitant medical condition that precludes intracerebroventricular administration, or use of anesthetics or immune suppression needed for study related procedures

Other inclusion and exclusion criteria apply.

Min Age: 3 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of NGN-401 | 52 Weeks
  Responders will be defined as participants who:
  * Attain a CGI-I score of ≤ 3 ("minimally improved");
  * and gain any one developmental milestone/skill from a list of 28, as captured through standardized video recordings and independently verified by blinded central raters.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Jordan, MD, Study Director — Neurogene Inc.
Locations (16):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nicklaus Children's Hospital Research Institute, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Montefiore Medical Center, New York, New York
  - UNC at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
- The Children's Hospital at Westmead, Sydney, New South Wales, Australia
- United Kingdom (2):
  - Royal Hospital for Children and Young People, Edinburgh
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ross PD, Gadalla KKE, Thomson SR, Selfridge J, Bahey NG, Benito J, Burstein SR, McMinn R, Bolon B, Hector RD, Cobb SR. Self-regulating gene therapy ameliorates phenotypes and overcomes gene dosage sensitivity in a mouse model of Rett syndrome. Sci Transl Med. 2025 Apr 2;17(792):eadq3614. doi: 10.1126/scitranslmed.adq3614. Epub 2025 Apr 2. PMID 40173263
- [Derived] Jagadeeswaran I, Oh J, Sinnett SE. Preclinical Milestones in MECP2 Gene Transfer for Treating Rett Syndrome. Dev Neurosci. 2025;47(2):147-156. doi: 10.1159/000539267. Epub 2024 May 9. PMID 38723617